CLINICAL TRIAL: NCT05605977
Title: Effectiveness of Home-based Visual-motor Training Programs on At-risk Kindergarteners
Brief Title: Home-based Visual-motor Training Program on Kindergarteners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-110-065
Record Dates: First submitted 2022-10-23; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-08

CONDITIONS: Developmental Delay; Preterm Children
Keywords: visual motor, kindergarten children, developmental delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: pretest-posttest control group design
Who Masked: Outcomes Assessor
Masking Description: The assessors are blinded to the assigned group of participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): regular early intervention
- Traditional visual-motor training program (Experimental): traditional visual-motor training program plus regular early intervention
  Interventions: Behavioral: Traditional visual-motor training program
- Computerized visual-motor training program (Experimental): computerized visual-motor training program plus regular early intervention
  Interventions: Behavioral: Computerized visual-motor training program

INTERVENTIONS:
Behavioral: Traditional visual-motor training program — Traditional visual-motor program includes play and paper-and-pencil activities
  Arms: Traditional visual-motor training program
Behavioral: Computerized visual-motor training program — Computerized visual-motor training program includes tablet visual-motor games
  Arms: Computerized visual-motor training program

SUMMARY:
The study aims to investigate the feasibility and effectiveness of the traditional and computerized home-based visual-motor training programs on at-risk kindergarteners.

DETAILED DESCRIPTION:
The purpose of this project is to investigate the feasibility and effectiveness of home-based traditional visual-motor activities and tablet games on fine motor, visual perception, visuo-motor integration, handwriting performance, and adaptive behaviors of at-risk kindergarteners. At-risk kindergarteners will be randomized into the three groups: control, traditional, and tablet groups. In addition to regular early intervention, children in the traditional and tablet group will receive home-based visuo-motor training program with their parents. Children in the control group will only receive regular intervention during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Either visual perception or fine motor score below the norm average
2. can follow instruction and complete the entire tests

Exclusion Criteria:

1. Visual or hearing problems that cannot be corrected to be normal
2. A diagnosis of significant neurological, muscular, and skeletal system disorders (e.g., Cerebral palsy)
3. A diagnosis of moderate or severe intellectual disabilities
4. Taking medication to control seizure or improve learning abilities

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
the Test of Visual Perceptual Skills-Fourth Edition (TVPS-4) | baseline, after 12 weeks
  the change of visual-perceptual skills
the Bruininks-Oseretsky Test of Motor Proficiency-Second Edition (BOT-2) | baseline, after 12 weeks
  the change of fine motor skills
the Chinese Handwriting Test | baseline, after 12 weeks
  the change of the Chinese handwriting performance

SECONDARY OUTCOMES:
The Berry-Buktenica Developmental Test of Visual-Motor Integration- Forth Edition (VMI) | baseline, after 12 weeks
  the change of VMI
the Vineland Adaptive Behavior Scales - Third Edition - Chinese Version (VABS-3-C) (Parents/Caregivers Edition)adaptive behavior | baseline, after 12 weeks
  the change of adaptive behavior
the test of Visual Perception of Chinese Characters | baseline, after 12 weeks
  The change of visual perception of Chinese characters
the Game Questionnaire | through study completion, an average of one week
  The questionnaire is designed to measure the difficulty, participation, and liking level of playing the training games using 5-point Likert scale from parental view after the completion of the games.
Parental Feedback Questionnaire | after 12 weeks
  The questionnaire consists of a few open-ended questions which are designed to realize parental experience of participating the home-based visual-motor training program.

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Shwu Hwang, ScD, Principal Investigator — National Cheng Kung University

IPD SHARING:
Plan to Share IPD: No
IPD are to be shared with other researchers

REFERENCES:
- [Background] Chen YN, Lin CK, Wei TS, Liu CH, Wuang YP. The effectiveness of multimedia visual perceptual training groups for the preschool children with developmental delay. Res Dev Disabil. 2013 Dec;34(12):4447-54. doi: 10.1016/j.ridd.2013.09.023. Epub 2013 Oct 11. PMID 24120756
- [Background] Lin LY, Cherng RJ, Chen YJ. Effect of Touch Screen Tablet Use on Fine Motor Development of Young Children. Phys Occup Ther Pediatr. 2017 Oct 20;37(5):457-467. doi: 10.1080/01942638.2016.1255290. Epub 2017 Jan 10. PMID 28071977
- [Background] Poon KW, Li-Tsang CW, Weiss TP, Rosenblum S. The effect of a computerized visual perception and visual-motor integration training program on improving Chinese handwriting of children with handwriting difficulties. Res Dev Disabil. 2010 Nov-Dec;31(6):1552-60. doi: 10.1016/j.ridd.2010.06.001. PMID 20621444